CLINICAL TRIAL: NCT05415982
Title: Diet Induced Ketosis for Patients With Posttraumatic Stress Disorder (PTSD), a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ketosis PTSD
Record Dates: First submitted 2022-03-23; First posted 2022-06-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): Ketogenic Diet every day for 4 weeks
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — The intervention is a ketogenic diet based on high-fat ketogenic meals prepared by the study participants, complemented with ketogenic food products from Natural Ketosis and Vitaflo. Exogenous ketones are provided by Audacious Nutrition. The macronutrient composition of the ketogenic diet given approx.: Fat 87 E%, Carbohydrate 3 E%, Protein 10 E%,

SUMMARY:
Many patients suffering from posttraumatic stress disorder (PTSD) are resistant to established treatment consisting of psychotherapy. Patients often go years with this debilitating disorder without experiencing sufficient improvement. Approximately 1/3 of patients will drop out of treatment because of psychological burden and overactivation. A novel ketogenic diet treatment could amend established treatment, and potentially upregulate the threshold for exciting neurons in dysfunctional brain regions, mediated through various mechanisms. This may reduce PTSD symptoms, and thus enabling patients to respond to psychological treatment without getting overactivated and unable to process trauma. The purpose of this study is to investigate whether it is possible to carry out a ketogenic diet therapy for patients with PTSD for four weeks.

DETAILED DESCRIPTION:
The study aims to include 10 PTSD patients. If a participant drops out of the study, or if the study is otherwise terminated for a participant, another patient will be recruited until 10 have completed the study. The primary objectives of this feasibility study are to investigate if it is possbile to carry out a ketogenic diet therapy for patients with PTSD for 4 weeks, and systematically gain insight in all challenges relating to these objectives. The participants will follow a ketogenic diet for 4 weeks, and they are asked to self report daily on results from finger pricking blood measurements (glucose and betahydroxybutyrate (BHB)) to establish they are in a ketogenic state and are compliant to diet. Participants will also report food intake and side effects daily to be evaluated by the principal investigator. Participants are further asked to specify and elaborate on which adverse effects or other reasons as to why it is challenging to follow the study diet and/or procedures. The study lacks in power to statistically evaluate if ketosis has any effect on PTSD symptoms, however this secondary objective will be preliminary evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years
* Diagnosed with posttraumatic stress disorder (PTSD)
* Understand and speak Scandinavian language

Exclusion Criteria:

* Body Mass Index < 18
* Metabolic disorders contraindicating a ketogenic diet
* Dysregulated Diabetes Mellitus
* Medicated for elevated triglycerides
* Pancreas, kidney or liver disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Recruitment | 25 weeks
  How many patients can be included in the intervention group (percent out of all eligible patients during the inclusion period)
Completing the intervention | 4 weeks
  How many patients complete the intervention of four weeks (percent out of all included patients) Completion is defined as adherence to the intervention daily for four weeks.
Maintaining ketosis | 4 weeks
  Could ketosis (mean b-BHB ≥ 0,5 mmol/L out of three daily measurements) be maintained for the duration of intervention (percent out of intervention days since ketosis first was obtained)
Adverse reactions related to the ketogenic treatment | 4 weeks
  The occurrence of adverse reactions (percent of days with adverse reactions during intervention)

SECONDARY OUTCOMES:
Assessment of severity of PTSD symptoms | 4 weeks
  Change in PTSD Checklist for DSM-5 scale (PCL-5). 20 part item, 0-4 likert scale. Minimum value 0, maximum value 80 (Lower score is better)
Measure of Health-Related Quality of Life | 4 weeks
  Change in RAND 36-Item Health Survey 1.0 (RAND-36) - Scale is converted to numerical values for physical and mental health (each item is scored on a 0 to 100 range, so that the lowest and highest score are 0 and 100, respectively). Items in the same scale are averaged together to create 8 scale scores. A higher score defines a more faborable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Furuholmen-Jenssen, Student, Principal Investigator — University of Copenhagen; Jens R Andersen, MD, MPA, Study Director — University of Copenhagen
Locations (1):
- Søndre Oslo Distriktspsykiatriske Senter (DPS), Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards MGP, Furuholmen-Jenssen T, Soegaard EGI, Thapa SB, Andersen JR. Exploring diet-induced ketosis with exogenous ketone supplementation as a potential intervention in post-traumatic stress disorder: a feasibility study. Front Nutr. 2024 Oct 31;11:1406366. doi: 10.3389/fnut.2024.1406366. eCollection 2024. PMID 39588043